### Informed Consent 30 July 2025

Feasibility of an RCT Examining
Effects of Active Plant Engagement
on
College Student Well-Being and
Performance

# Consent to Participate in a Research Study Colorado State University

## TITLE OF STUDY: Feasibility of an RCT Examining Effects of Active Plant Engagement on College Student Well-Being and Performance

### PRINCIPAL INVESTIGATOR:

Kaigang Li, Ph.D.
Department of Health and Exercise Science
Colorado State University
Fort Collins
CO 80523-1582

Telephone: (970) 491-7253

Email: Kaigang.Li@colostate.edu

### **INVITATION TO PARTICIPATE**

You are invited to participate in a research study about how caring for plants may affect college students' mental health and academic performance. Your participation is voluntary.

#### WHY IS THIS STUDY BEING DONE?

This study aims to:

- Compare how caring for plants at home versus on campus affects stress and academic habits
- Understand if active plant care is more beneficial than passive exposure

### **HOW MANY PEOPLE WILL PARTICIPATE?**

We plan to enroll ~90 CSU students (~30 in each group).

### WHAT WILL HAPPEN IF I PARTICIPATE?

If you agree:

- 1. You'll be randomly assigned to one of three groups:
  - o **Group 1:** Complete surveys only (no plants) o
    - Group 2: Care for plants on campus + surveys
  - Group 3: Care for plants at home + surveys 2.
     Complete 4 online surveys (15-20 mins each) over 16 weeks 3. If in Groups 2 or 3:
  - Receive 1-2 easy-care plants Do weekly care tasks (watering, pruning) Take monthly plant photos

### **HOW LONG WILL I PARTICIPATE?**

- 16 weeks (one semester)
- The last survey (Week 16) is optional

### ARE THERE RISKS?

This study involves minimal risk. Potential risks include minor plant allergies, psychological stress (e.g., if plants do not thrive), and time commitment (approximately 30 minutes per week). *To mitigate these risks:* 

- Allergies: Only hypoallergenic plants will be provided.
- Psychological Distress: You could contact CSU Mental Health Services at (970) 4917121 as needed.
- Emergency Protocol: In the event of a severe reaction, please contact the CSU Health and Medical Center at (970) 491-7121.

## **Are There Any Benefits from Taking Part in the Study?** This study is not designed to benefit you directly.

### Will I Receive Compensation?

You will be paid for being in this research study. You will receive up to \$40 for completing the surveys. In addition, all participants will receive free plants after the study: Group 1 will receive new plants, while Groups 2 and 3 will keep the plants assigned to them during the study.

### WHO WILL SEE THE INFORMATION THAT I GIVE?

We will keep all the research records that identify you private, to the extent allowed by law. Your information will be combined with information from other people taking part in the study. When we write about the study to share with other researchers, we will write about the combined information we have gathered. You will not be identified in these written materials. We may publish the results of this study; however, we will keep your name and other identifying information private. We may be asked to share the research files with the CSU Institutional Review Board ethics committee for auditing purposes. Your identity/record of receiving compensation (NOT your data) may be made available to CSU officials for financial audits.

### **CLINICALTRIALS.GOV REGISTRATION**

A description of this clinical trial will be available on http://www.ClincialTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

### CAN MY TAKING PART IN THE STUDY END EARLY?

Your participation in the study may end early if there are any complications or signs of abnormal response to plants during the study.

### WHAT IF I CHANGE MY MIND?

You may quit anytime without penalty. You will be compensated for the surveys you complete.

### **FUTURE USE OF DATA COLLECTED**

| It is possible that we may want to use the data collected during this study for future studies. We will keep private all research records that identify you (to the extent allowed by law) for both current and future use (please refer to the section, "WHO WILL SEE THE INFORMATION THAT |
|---|
| I GIVE" for more information regarding privacy). Choose only one of the following: |
| Please scroll down and provide your initials and signature in the boxes below the consent. |
| I give permission for the use of data collected for the current study only. |
| (your initials) |
| Please scroll down and provide your initials and signature in the boxes below the consent. |
| I give permission for the use of data collected for the current study as well as for future |
| studies. |
| (your initials) |
| () •, |

### WHO CAN ANSWER MY QUESTIONS?

- Study questions: Dr. Li at <a href="mailto:Kaigang.Li@colostate.edu">Kaigang.Li@colostate.edu</a> or (970) 491-7253
- Rights questions: CSU IRB at CSU IRB@colostate.edu or 970-491-1553

### YOUR CONSENT

By signing, you confirm:

- √ Your participation is voluntary
- √ You're ≥18 years old
- ✓ You have NO concurrent participation in similar wellness/mental health studies
- √ You have NO current plant-growing activities
- √ You are NOT allergic to hypoallergenic plants (e.g., pothos, snake plants, peace lilies)

Your signature acknowledges that you have read the information stated and willingly sign this consent form. Your signature also acknowledges that you have received, on the date signed, a copy of this document containing 3 pages.

| Signature of person agreeing to take part in the study | Date | _ |
|-----------------------------------------------------------|-------------|---|
| Printed name of person agreeing to take part in the study | Time of Day | _ |
| Name of person providing information to participant | Date | |
| Signature of Research Staff | | |